CLINICAL TRIAL: NCT02842229
Title: Retrospective Study to Determine Final Geriatric Assessment in Haematology (GAH) Score as a Tool for Predicting Tolerance to Treatment in Elderly Patients (≥ 65 Years) With Haematologic Neoplasms
Brief Title: A Study to Determine Final Geriatric Assessment in Haematology (GAH) Score as a Tool for Predicting Tolerance to Treatment in Elderly Patients (≥ 65 Years) With Haematologic Neoplasms
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL-GAH-2016-01
Record Dates: First submitted 2016-06-21; First posted 2016-07-22 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Myelodysplastic Syndromes; Leukemia Myeloid Acute; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: Myelodysplastic Syndromes; Leukemia Myeloid Acute; Multiple Myeloma; Leukemia, Lymphocytic, Chronic; Elderly Patients; Haematological malignancy; Elderly; Health Status; Scale validation; Retrospective
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Haematologic Neoplasms: Patients with Myelodysplastic Syndromes (MDS), any IPSS (International Prognostic Scoring System) risk, or Acute Myeloid Leukemia (AML) who participated in the Geriatric Assessment in Haematology (GAH) study(CEL-GAH-2011-01).
  Patients with Multiple Myeloma (MM), symptomatic or asymptomatic who participated in the Geriatric Assessment in Haematology (GAH) study (CEL-GAH-2011-01).
  Patients with Chronic Lymphocytic Leukemia who participated in the Geriatric Assessment in Haematology (GAH) study (CEL-GAH-2011-01).

SUMMARY:
This is a post-authorization, retrospective multicentre observational nationwide study (PAS-OD). It will be conducted by reviewing medical records and database of patients who participated in the validation of the psychometric properties of the GAH study (CEL-GAH-2011-01). In all cases, only data prior to the start date of the study will be collected to ensure its retrospective nature, thereby reflecting routine clinical practice and non-interference in the physician's clinical practice

DETAILED DESCRIPTION:
Patients over 65 are the most prevalent population in oncological clinical practice. It is also expected that this group of patients will increase significantly in the coming decades as a result of increased life expectancy and the aging population.

Overall, the population is aging and this aging is accompanied by an increase in the prevalence and incidence of age-related diseases, such as cancer. So much so that approximately 60% of new cancer cases and 70% of the overall cancer mortality occurs in patients aged 65 and over.

Despite the high incidence of cancer in the elderly and its peculiarities as opposed to young patients, from the point of view of health, the management of elderly patients is especially complex because there are few data on the evaluation and treatment thereof. Often, older patients are underrepresented in clinical trials and treatment guidelines, resulting in a population that is undertreated or at greater risk of suffering treatment-related toxicities.

In this respect, both the National Comprehensive Cancer Network (NCCN) and the International Society of Geriatric Oncology (SIOG, its acronym in Spanish) agree that age should not be an impediment to treat these diseases. Optimal management requires strategies specifically directed to the clinical and biological characteristics of this type of patient and they recommend an appropriate assessment of the patient as part of a safe and effective approach to haematological malignancies in the elderly.

There is scientific basis supporting the need for the elderly patient with cancer who will receive a particular treatment to be specifically assessed by means of a comprehensive geriatric assessment (CGA). Geriatric assessment is essential since it is a tool that integrates all aspects of the patient's life that could affect the course of the disease and response to treatment, such as functional status, comorbidities, cognitive, emotional or nutritional status and social environment. In addition, the CGA is a tool to identify the possible presence of fragility, characterized by a decrease in physiological reserves that conditions a lower response to stress and is associated with a lower risk of disability and increased morbidity and mortality.

Although currently it is assumed that chronological age is not synonymous with biological age, the decision on cancer treatment often falls on the subjective assessment of the physician, as few healthcare centres are performing comprehensive geriatric assessment in the oncology setting. Although various tools have been developed for this purpose, they have not been incorporated into routine clinical practice due to the time required, their length and the resources needed to gather information.

Therefore, there remains a need to find a scale for comprehensive assessment of the health status of elderly patients (≥ 65 years) with haematologic malignancies that incorporates the essential dimensions of the geriatric assessment, with the same precision of valid tools currently available, and that is simple, straightforward and easy to apply, so that it can be used in daily practice and assist to make clinical decisions objectively.

It was hypothesized that a simplified geriatric assessment could be a better tool for assessing elderly patients, instead of considering only age or subjective clinical impression, when deciding whether or not to prescribe active treatment. Such a tool would represent the real and multidimensional nature of aging, which is associated with an increased incidence of chronic diseases and geriatric syndromes with consequences on vulnerability and patient survival.

As described above, Bonanad et al. designed and developed a new comprehensive assessment scale aimed at elderly patients (≥ 65 years) diagnosed with haematological diseases [myelodysplastic syndrome (MDS) or Acute myeloid leukemia (AML), multiple myeloma (MM) and chronic lymphocytic leukemia (LLC)], the Geriatric Assessment in Haematology (GAH). The purpose of this scale is to help doctors identify objectively and reliably those elderly patients with haematological diseases who are eligible for intensive treatment versus those who are most vulnerable.

The GAH scale is a tool of 30 items grouped into eight relevant dimensions of geriatric assessment, which include:

1. Number of drugs: Polypharmacy has been associated with adverse effects related to frailty, disability, mortality and falls in the elderly, and it may be more frequent in elderly patients with cancer.
2. Gait velocity: Determining the time taken to walk four meters at a normal pace is a method of assessing gait velocity that is widely used in the literature due to its simplicity, speed and reliability. There is sufficient evidence to consider walking speed as a strong and consistent predictor of adverse outcomes in older patients, and its use as a single item has proven to be at least as sensitive as compound instruments in predicting most of these results long-term.
3. Mood: We propose as a screening test for depression a single item extracted from the Center for Epidemiologic Studies Depression Scale (CES-D), widely used for its validity and reliability. This unique and simple measure of depression was shown to be strongly correlated with a clinical diagnosis of depression; it detects patients rarely or sometimes depressed and patients depressed occasionally or much of the time.
4. Activities of daily living: The assessment of functional status in older people should include assessment of so-called basic activities of daily living (ADLs), including the skills necessary for life such as dressing, grooming, bathing and feeding. ADL is a tool that has been used as a predictor of hospitalization and mortality in elderly patients.

   To develop the activities of daily living (ADL) of the GAH scale, items were selected from the Vulnerable Elders Survey (VES-13) with two additional questions.
5. Subjective health status: The patient rating his or her own health is another worthwhile parameter. This is why a self-rated health item was also selected, also included in the Vulnerable Elders Survey (VES-13). Recently it has been determined that this is a predictive parameter of functional impairment or death.
6. Nutrition: Nutritional deficit is a common serious problem in elderly patients, contributing significantly to morbidity and mortality associated with this group of people. To determine this dimension, some items were selected from the short version of the full questionnaire, Mini-Nutritional Assessment. This tool was developed and validated in representative samples of older patients worldwide and it identifies subjects at nutritional risk.
7. Mental State: To evaluate mental state, all the items were selected that make up the Short Portable Mental Status Questionnaire (SPMSQ). It is designed and validated to assess four aspects of intellectual functioning: short and long-term memory, orientation, information on daily events and computing ability. It has been observed that cognitive impairment is also an independent predictor of mortality and the end of chemotherapy.
8. Comorbidity: Six variables of comorbidity and habits were considered (diabetes mellitus, cancer, lung disease, heart failure, smoking), drawn from the Prognostic Index for 4-year Mortality in Older Adults.

The final score of the GAH scale has not yet been defined. At present, for purely exploratory purposes, each of the dimensions was assigned a dichotomous score (0 or 1), generating a provisional score ranging from 0 (best possible health status) to 8 (worst health status). The recently published study showed that the GAH scale is a measuring instrument that meets the expected psychometric properties (feasibility, ceiling-floor effect, reliability and validity) for a tool to determine health status in elderly patients with haematological diseases. Also, it has been determined that this scale is sensitive to change <pending (reference short report)>, since it is able to detect changes in the health status of patients after a certain time and is able to predict survival in this patient group.

This study aims to determine the weights of each of the dimensions of the GAH scale, as well as cut-off points for the final score of the scale that will be used to predict treatment tolerability in elderly patients diagnosed with MDS/ AML, MM or CLL (chronic lymphocytic leukemia).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were participating in the GAH study (CEL-GAH-2011-01).
* Patients who have been scheduled to start treatment at a date less than three months after completion of the GAH (CEL-GAH-2011-01) scale in one of these visits: baseline, test-retest or sensitivity to change.
* Patients who give informed consent to participate in the study as long as such consent is possible.

Exclusion Criteria:

• Not applicable

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: At least 80 patients will be included who participated in the Geriatric Assessment in Haematology (GAH) study (CEL-GAH-2011-01), who are scheduled to start treatment less than three months after completion of the GAH assessment (basal, test-retest or sensitivity to change) and who give their informed consent to data collection as long as such consent is possible.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Assessment of the tolerability of the treatment administered | Up to approximately 4 months
  Number of patients, which suspend or modify treatment due to toxicity
The score of number of drugs on the Geriatric Assessment in Haematology (GAH) scale | Up to approximately 4 months
  Determination of number of drugs that patients were taken.
The time of gait velocity on the Geriatric Assessment in Haematology (GAH) scale | Up to approximately 4 months
  To determine the time taken to walk four meters at a normal pace.
The score of activities of daily living on th Geriatric Assessment in Haematology (GAH) scale | Up to approximately 4 months
  Assessment of so-called basic activities of daily living (ADLs), including the skills necessary for life such as dressing, grooming, bathing and feeding
The score of subjective health status on the Geriatric Assessment in Haematology (GAH) scale | Up to approximately 4 months
  The patient rating his or her own health
The score of nutrition on the Geriatric Assessment in Haematology (GAH) scale | Up to approximately 4 months
  To determine nutritional deficit
The score of mental State on the Geriatric Assessment in Haematology (GAH) scale | Up to approximately 4 months
  To evaluate mental state
The score of comorbidity on the Geriatric Assessment in Haematology (GAH) scale | Up to approximately 4 months
  Six variables of comorbidity and habits were considered (diabetes mellitus, cancer, lung disease, heart failure, smoking)

SECONDARY OUTCOMES:
Therapeutic approach according to clinical judgment | Up to approximately 4 months
  Number of patients that due to their fragility, the physician decided to modify the planned start treatment.
Discontinuation of the planned treatment due to toxicity | Up to approximately 4 months
  Percentage of patients who discontinued the planned treatment due to toxicity
Modification of the planned treatment regimen due to toxicity | Up to approximately 4 months
  Percentage of patients who modified the planned treatment regimen due to toxicity
Percentage of patients with toxicity | Up to approximately 4 months
  Percentage of patients who suspend or amend the treatment regimen due toxicity
Number of participants visit to hospital as a result of toxicity | Up to approximately 4 months
  Number of patients who were admitted to hospital as a result of toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Marta Duran, PhD, Study Director — Celgene Corporation
Locations (15):
- Spain (15):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Durán I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - C.H. Universitario A Coruña, A Coruña, La Coruña
  - C. H. Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Ntra. Sra. La Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital La Ribera, Alzira, Valencia
  - Hospital Vall d' Hebrón, Barcelona
  - Hospital U. Gregorio Marañón, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital de Segovia, Segovia
  - Hospital La Fe, Valencia
  - Hospital Txagorritxu, Vitoria-Gasteiz, Álava